CLINICAL TRIAL: NCT03316001
Title: Mesenteric Panniculitis : Review of Consecutive Abdominal MDCT Examinations With a Matched-pair Analysis
Acronym: MP - Cancer
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: 2016Ao002
Record Dates: First submitted 2017-10-17; First posted 2017-10-20 (Actual); Last update posted 2017-10-20 (Actual); Status verified 2017-10

CONDITIONS: Mesenteric Panniculitis
MeSH Terms: conditions — Panniculitis, Peritoneal

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cases: patients with a CT scan from January to August 2008 for which mesenteric panniculitis was diagnosed
  Interventions: Other: Review of multidetector row computed tomography scans
- controls: patients with a CT scan from January to August 2008 for which mesenteric panniculitis wasn't diagnosed and matched by gender and age with "cases" patients
  Interventions: Other: Review of multidetector row computed tomography scans

INTERVENTIONS:
Other: Review of multidetector row computed tomography scans — multidetector row computed tomography scans

SUMMARY:
Mesenteric panniculitis is a benign inflammatory condition that involves the adipose tissue of the intestinal mesentery. Clinical manifestations are uncommon, non specific and atypical. Mesenteric panniculitis is thus most often an incidental finding during an investigation for other reason, mostly on computed tomography scans. The rate of malignancy in patients with mesenteric panniculitis, especially urogenital and gastrointestinal adenocarcinomas or lymphomas, has been reported to be as high, thus suggesting that there may be a relationship between mesenteric panniculitis and progression of an underlying malignancy or the risk of a future malignancy.

DETAILED DESCRIPTION:
The aim was:

to estimate the prevalence of mesenteric panniculitis. to study relationship between mesenteric panniculitis and malignancy. to investigate the 5-year outcome of patients with mesenteric panniculitis for the development of malignancy.

ELIGIBILITY:
inclusion criteria:

* Patients with a CT scan from January to August 2008
* Patients with diagnosis of mesenteric panniculitis on CT scan

exclusion criteria:

* Patients with disease that may cause mesenteric infiltration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a CT scan from January to August 2008 for which mesenteric panniculitis was diagnosed
Sampling Method: Non-Probability Sample
Enrollment: 288 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
mesenteric panniculitis | Day 0
  mesenteric panniculitis is identified on the basis on the presence of three of the following 5 signs on CT scan:
  * higher attenuation of the fat of the root of the small bowel mesentery,
  * a pseudo mass smoothly displacing neighboring structures with a hyperdense pseudocapsule surrounding the mesenteric fat,
  * lymph nodes within the fatty pseudo mass and
  * a hypodense halo around the nodes and the blood vessels

REFERENCES:
- [Background] Protin-Catteau L, Thiefin G, Barbe C, Jolly D, Soyer P, Hoeffel C. Mesenteric panniculitis: review of consecutive abdominal MDCT examinations with a matched-pair analysis. Acta Radiol. 2016 Dec;57(12):1438-1444. doi: 10.1177/0284185116629829. Epub 2016 Jul 19. PMID 26868171